CLINICAL TRIAL: NCT06667349
Title: Ticagrelor Intervention to Suppress Stent Thrombosis and Acute MI Risk (TISSARA) Trial: An LMIC Health System Initiative in the World's Busiest Primary PCI Center
Brief Title: TISSARA Trial: Ticagrelor Intervention to Reduce Stent Thrombosis and Acute MI Risk
Acronym: TISSARA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Cardiovascular Diseases, Pakistan (Other)
Responsible Party: Principal Investigator, Professor Abdul Hakeem, Professor Abdul Hakeem MD FACC FSCAI FASE, National Institute of Cardiovascular Diseases, Pakistan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NICVD IRB-40/2023
Record Dates: First submitted 2024-09-28; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; Stent Thrombosis; Antiplatelet Agents
Keywords: clinical trial; STEMI; stent thrombosis; ticagrelor; clopidogrel; health care intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Ticagrelor

STUDY DESIGN:
Intervention Model Description: 1727
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tiacgrelor (Tissara) 90 mg pod BID (Experimental): Ticagrelor 90 mg bid give for atleast two weeks and ideally upto a month
  Interventions: Drug: Ticagrelor
- standard arm clopidogrel 75 mg qday (Active Comparator)
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor 90 mg PO BID given for atleast two weeks following primary PCI
  Other Names: Brilinta

SUMMARY:
Stent thrombosis (ST) remains a critical complication following primary percutaneous coronary intervention (PPCI) in patients with ST-elevation myocardial infarction (STEMI). At the National Institute of Cardiovascular Diseases in Karachi-recognized as the world's busiest PPCI center-reported rates of ST range from 4% to 6%. In response to this pressing issue, the health system has implemented a new two-week post-PCI regimen featuring ticagrelor, aimed at enhancing patient outcomes and reducing the risk of stent-related complications.

The TISSARA Trial is designed to rigorously assess the effectiveness of this intervention on cardiovascular outcomes in STEMI patients.

Between August, 2023 and March 2024, a total of 1,773 patients were enrolled in the trial, with 970 patients discharged on Tissara (Ticagrelor) (Ferozsons laboratories Ltd, Lahore, Pakistan) (TG) and 803 patients receiving clopidogrel (CG) following their primary PCI procedures. Each group was carefully monitored for a duration of three months to evaluate the incidence of stent thrombosis and other relevant cardiovascular events. The primary endpoint of this trial is the occurrence of stent thrombosis within the follow-up period, providing critical insights into the safety and efficacy of the ticagrelor regimen in this high-risk population.

This comprehensive approach aims to contribute valuable data that may influence future treatment protocols and improve the standard of care for patients undergoing PCI in similar healthcare settings.

DETAILED DESCRIPTION:
The TISSARA Trial aims to compare the incidence rates of stent thrombosis (ST) and major adverse cardiovascular events (MACE) among patients receiving ticagrelor therapy versus those treated with conventional clopidogrel therapy following primary percutaneous coronary intervention (PPCI) f or ST elevation myocardial infarction at NICVD, Karachi, Pakistan.

Study Cohorts:

* Ticagrelor Cohort: Comprises consecutive patients receiving ticagrelor as part of the dual antiplatelet therapy (DAPT) regimen mandated for a minimum of two weeks post PPCI.
* Clopidogrel Cohort: Included patients who received clopidogrel as part of the conventional DAPT protocol.

Selection Criteria:

• All consecutive patients presenting with ST-elevation myocardial infarction (STEMI) and undergoing primary PCI with drug-eluting stents (DES).

Exclusion Criteria:

* Patients who underwent plain old balloon angioplasty (POBA) or left heart catheterization (LHC) only.
* Patients who declined to provide consent.
* Patient with high bleeding risk
* Prior history of IC hemorrhage
* Prior CVA within past one year
* On oral anticoagulant Study Variables and Operational Definitions
* ST-Elevation Myocardial Infarction (STEMI): Diagnosis based on at least two of the following criteria:

  * Typical chest pain lasting more than 20 minutes, characterized by retrosternal pain radiating to the left arm or shoulder, worsening with exertion or emotional stress, and alleviated by rest or nitroglycerin.
  * New ST elevation in at least two contiguous leads: greater than 2 mm in men or greater than 1 mm in women in leads V2 to V3, and/or greater than 1 mm in other contiguous chest leads or limb leads.
* Primary PCI: The strategy of directly taking a STEMI patient to the cardiac catheterization laboratory for mechanical revascularization via balloon angioplasty and coronary stenting.
* Stent Thrombosis:

  * Definite Stent Thrombosis: Confirmed by angiographic or pathological evidence of partial or total thrombotic occlusion within the peri-stent area, along with acute ischemic symptoms, ischemic ECG changes, or elevated cardiac biomarkers.
  * Probable Stent Thrombosis: Unexplained death within 30 days of stent implantation or myocardial infarction related to documented acute ischemia in the stented territory, without angiographic confirmation of stent thrombosis.
  * Possible Stent Thrombosis: Unexplained death occurring beyond 30 days.
  * Early Stent Thrombosis: Occurs within 24 hours post-PCI.
  * Subacute Stent Thrombosis: Occurs from 24 hours to 30 days post-PCI.
* Major Adverse Cardiovascular Events (MACE): Defined as a composite of:

  * All-cause mortality
  * Cardiovascular mortality
  * Myocardial infarction (with or without revascularization)
  * Unplanned hospitalization due to heart failure
  * Stroke or cerebrovascular events Data Collection Procedure The study was conducted after receiving approval from the ethical review committee of NICVD, Karachi. Verbal informed consent was obtained from all participants, ensuring confidentiality. Patients presenting with STEMI who underwent primary PCI with second-generation DES were included. Data on demographic characteristics, financial status, treatment compliance, complications, hospitalizations, and emergency room visits were collected using a structured questionnaire. The collected data were securely stored and accessible to the primary investigators and co-investigators. Patients were followed up at 15 days and one month in the outpatient clinic to assess medication compliance, side effects, and bleeding.

ELIGIBILITY:
Inclusion Criteria: consecutive patients presenting with ST-elevation myocardial infarction (STEMI) and undergoing primary PCI with drug-eluting stents (DES).

-

Exclusion Criteria:

* Patients who underwent plain old balloon angioplasty (POBA) or left heart catheterization (LHC) only.

  * Patients who declined to provide consent.
  * Patient with high bleeding risk
  * Prior history of IC hemorrhage
  * Prior CVA within past one year
  * On oral anticoagulant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1727 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2024-03-03 (Actual); Study Completion 2024-06-16 (Actual)

PRIMARY OUTCOMES:
Stent Thrombosis | Stent thrombosis occurring 24 hours to 30 DAYS
  A. Definite Stent Thrombosis: Angiographic or pathological confirmation of partial or total thrombotic occlusion within the peri-stent region and at least one of the following additional criteria: Acute ischemic symptoms Ischemic electrocardiogram changes Elevated cardiac biomarkers
  B. Probable Stent Thrombosis:
  Any unexplained death <30 days of stent implantation Any myocardial infarction related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause C. Possible Stent Thrombosis: Any unexplained death beyond 30 days D. Early Stent Thrombosis: Stent thrombosis occurring within 24 hours E. Subacute Stent Thrombosis: Stent thrombosis occurring 24 hours to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Hakeem, MD, Principal Investigator — National Institute of Cardiovascular Diseases
Locations (1):
- National Institute of Cardiovascular Diseases, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Kumar R, Ammar A, Saghir T, Sial JA, Shah JA, Kumar A, Shaikh AH, Achakzai AS, Qamar N, Karim M. Incidence, Predictors, and Outcomes of Acute and Sub-acute Stent Thrombosis after Emergency Percutaneous Coronary Revascularization with Drug-Eluting Stents: A Prospective Observational Study. Glob Heart. 2022 Mar 30;17(1):24. doi: 10.5334/gh.1112. eCollection 2022. PMID 35586746
- [Background] Schulz S, Schuster T, Mehilli J, Byrne RA, Ellert J, Massberg S, Goedel J, Bruskina O, Ulm K, Schomig A, Kastrati A. Stent thrombosis after drug-eluting stent implantation: incidence, timing, and relation to discontinuation of clopidogrel therapy over a 4-year period. Eur Heart J. 2009 Nov;30(22):2714-21. doi: 10.1093/eurheartj/ehp275. Epub 2009 Jul 11. PMID 19596658
- [Background] Dubey G, Verma SK, Bahl VK. Primary percutaneous coronary intervention for acute ST elevation myocardial infarction: Outcomes and determinants of outcomes: A tertiary care center study from North India. Indian Heart J. 2017 May-Jun;69(3):294-298. doi: 10.1016/j.ihj.2016.11.322. Epub 2016 Nov 30. PMID 28648416